CLINICAL TRIAL: NCT01884766
Title: Prospective Study on Copeptin in Childhood Epilepsy
Brief Title: Copeptin in Childhood Epilepsy
Acronym: EpiCop
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University Children's Hospital Basel (Other)
Responsible Party: Sponsor
Other Study IDs: EKBB 352/12
Record Dates: First submitted 2013-05-10; First posted 2013-06-24 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Epilepsy; Febrile Seizures; Children
MeSH Terms: conditions — Epilepsy; Seizures, Febrile

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Epilepsy: All kind of epilepsy, including febrile seizures
- Control: children without seizures at presentation in the emergency but fever due to banal infections

SUMMARY:
In many fields of medicine, except seizure disorders, blood biomarkers have captured an integrated part of diagnostic decision making, including copeptin, the surrogate marker of vasopressin release. There are strong arguments to hypothesize circulating copeptin is elevated in epilepsy, especially in generalized seizures such as fever seizures (FS), and that copeptin is predictive for complexity and relapse at least in FS. Although long-term morbidity and mortality are both low in FS, there is high anxiety among parents because of a lack of criterions to identify children at risk for relapse. Copeptin may fill this gap by adding important diagnostic and prognostic information. Eventually, less children may receive needlessly over years fever drugs or anti-epileptic drugs.

DETAILED DESCRIPTION:
Background:

Copeptin is a surrogate marker of the pituitary-secreted nonapeptide arginine-vasopressin (AVP) and has gradually replaced AVP in several clinical studies largely due to its structural and methodological advantages. Copeptin is a marker of non-specific stress response, and has been suggested to have clinical implications in a variety of cardiovascular and non-cardiovascular conditions. However, up to now there are no data available on copeptin in seizure disorders, neither in adults nor in children.

Working hypotheses:

1. Circulating copeptin concentrations are increased after generalized seizures, including FS.
2. Copeptin is predictive for complexity and relapse in FS.

Specific aims:

1. to determine copeptin concentrations in children below six years after generalized seizures, either unrelated or related to fever (FS), and in control children below six years without seizures.
2. to compare copeptin concentrations with blood-gas parameters (including hydrogen ion concentration (pH), base deficiency, and carbon dioxide), lactate, sodium, chloride, C reactive protein (CRP), and prolactin.

ELIGIBILITY:
Inclusion Criteria epilepsy-cohort:

* All kind of seizures leading to presentation
* Age below 6 years

Inclusion Criteria control-cohort:

* Fever without seizures caused by banal infections
* Age below 6 years

Exclusion Criteria:

* No blood required for medical reasons

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children below six years presenting at the emergency unit of one tertiary university children's hospital
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Copeptin concentration in serum | at admission

SECONDARY OUTCOMES:
base excess in blood gas analysis | at admission
prolactin | at admission
duration of seizures | at admission
Short term relapse of seizures | 24 hours after first presentation
sodium concentration | at admission
osmolality | at admission
hydrogen ion activity in blood gas analysis | at admission
  hydrogen ion activity = pH

OTHER OUTCOMES:
number of repeated events of seizures | 12 month
  relapse of seizures within 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Sven Wellmann, MD, Principal Investigator — University Children's Hospital Basel, 4056 Basel, Switzerland
Locations (1):
- University Children's Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Stocklin B, Fouzas S, Schillinger P, Cayir S, Skendaj R, Ramser M, Weber P, Wellmann S. Copeptin as a serum biomarker of febrile seizures. PLoS One. 2015 Apr 20;10(4):e0124663. doi: 10.1371/journal.pone.0124663. eCollection 2015. PMID 25894585